CLINICAL TRIAL: NCT00250523
Title: Mathematical Modeling of the Acute Inflammatory Response Following Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dr Jason L Sperry, Professor of Surgery and Critical Care Medicine, National Institute of General Medical Sciences (NIGMS)
Other Study IDs: PRO 0801232; P50GM053789-09 (NIH)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Trauma; Critical Illness
Keywords: trauma; critical illness; injury
MeSH Terms: conditions — Wounds and Injuries; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For trauma injury cohort: The maximum blood volume collected over the 28 day period, if all samples are obtained, is approximately 90 cc. All standard precautions will be undertaken to assure minimal risk.
  Blood samples will be obtained for genetic analysis of inflammatory gene polymorphisms. We will collect whole blood, serum and white cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traumatic injury: ICU Patients with blunt or penetrating injury
- 2: Healthy volunteers

SUMMARY:
The purpose of this research study is to gather clinical and biologic information from severely injured patients to better understand and characterize the host response to injury and inflammation across several domains. This information may improve outcome prediction, improve clinical treatment of injured patients, and permit the construction of non-biologic computerized models of illness that can be utilized to represent the host response in future research efforts. This study is designed as the calibration of a mathematical model of this response with predictive capabilities.

The central hypothesis governing this study is that adaptive immune elements are crucial to determining the outcome of complex inflammatory scenarios. We propose to test these hypotheses in the following interrelated Specific Aims:

Specific Aim 1: To develop a robust mathematical model describing trauma/hemorrhage-induced inflammation in humans, its pathologic consequences, and possible therapies.

Specific Aim 2: To translate the mathematical model to humans and create software aimed at individualized clinical decision-making.

Specific Aim 3: To determine the prevalence of an IL-1 receptor-associated kinase (IRAK-1) variant haplotype located on the X-chromosome in an injured population, and to characterize differences in the pro-inflammatory response across gender, relative to the IRAK-1 haplotype.

Specific Aim 4: To determine if increased arginase activity previously observed in isolated peripheral blood mononuclear cells of trauma patients is a consequence of the presence of contaminating activated granulocytes or a particular subset of an arginase positive monocyte subset.

ELIGIBILITY:
Trauma patient cohort inclusion criteria:

* Present for treatment of their acute, blunt or penetrating injuries to the University of Pittsburgh Medical Center within 6 hours of injury
* Age greater than or equal to 18 years
* Intact cervical spinal cord
* Are admitted to the Intensive Care Unit

Trauma patient cohort exclusion criteria:

* Anticipated survival < 24 hrs
* Anticipated survival < 28 days due to pre-existing condition
* Traumatic Brain injury (GCS ≤8 after ICU admission) AND brain CT abnormality within 12 hr of injury
* Inability to obtain consent from the subject or their legally authorized representative.
* Pre-existing immunosuppression
* Transplant recipient
* Chronic high doses of steroids (>20 mg prednisone equivalents/day)
* Significant likelihood of high dose steroids (e.g. spinal cord injury)
* Oncolytic drug(s) therapy within the past 14 days
* Known HIV positive status and CD4 count < 200 cells/mm3
* Admission to the ICU primary for substance withdrawal.
* Inability to obtain 1st blood sample within 24 hours of injury.

Healthy volunteer cohort inclusion:

* Age greater than or equal to 18 years
* Weight > 110 pounds
* no recent illness or infection in the last two weeks
* no recent hospitalization or trauma in the last month

Healthy volunteer cohort exclusion:

* wt < 110 lbs
* infection or illness in the last two weeks
* Hospitalization or trauma in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited will consist of trauma patients and healthy volunteers:
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2003-02; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Multiple Organ Failure | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Sperry, MD, Principal Investigator — UPMC Department of Surgery/Critical Care Medicine
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No